CLINICAL TRIAL: NCT00907920
Title: Observational - Characterizing the Frequency and Spectrum of ALK Mutations in Neuroblastoma
Brief Title: Studying Tumor Samples From Young Patients With Neuroblastoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL09B1; NCI-2009-00501 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NB 2008-08 (Other: Children's Oncology Group)
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumor Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Correlative studies: Tumor DNA samples are examined by mutation analysis for germline and somatic mutations in the ALK tyrosine kinase domain. Samples are analyzed by whole genome amplification using polymerase chain reaction and then sequenced for DNA alterations in the entire ALK coding sequence. Samples are also examined for SNPs by polymorphism analysis. Exploratory multivariable analysis is performed to test for the prognostic ability of ALK mutations in the presence of other known prognostic variables (i.e., age, International Neuroblastoma Staging System stage, MYCN status, International Neuroblastoma Pathology Classification, and diploidy).
  A subset of tumor DNA samples from high-risk patients will be resequenced for DNA alterations to determine whether or not additional regions in ALK, outside of the tyrosine kinase domain, are prone to mutations and should be sequenced in a larger panel.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research study is looking at tumor samples from young patients with neuroblastoma. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer

DETAILED DESCRIPTION:
Study Subtype: Ancillary/Correlative Observational Study Model: Cohort Time Perspective: Retrospective Biospecimen Retention: Samples With DNA Biospecimen Description: Tissue Study Population Description: Patients previously enrolled on clinical trial COG-ANBL00B1 Sampling Method: Non-Probability Sample

PRIMARY OBJECTIVE:

I. To comprehensively identify and characterize the spectrum and frequency of mutations in ALK across all neuroblastoma disease subsets using methodologies that will be resource neutral to the Children's Oncology Group Neuroblastoma Nucleic Acids Bank.

SECONDARY OBJECTIVES:

I. To formulate genetic screening recommendations for newly diagnosed patients with or without a family history of neuroblastoma.

II. To identify the functionally relevant ALK mutations that can be pharmacologically inhibited.

III. To test for the prognostic capability of ALK alterations. IV. To determine the clinical significance of ALK mutations and/or genomic rearrangements by combining ALK mutation, amplification, and translocation data overall and within each neuroblastoma risk group and correlating this information with clinical phenotype (i.e., age, International Neuroblastoma Staging System stage, and International Neuroblastoma Pathology Classification); genetic factors (i.e., ploidy, MYCN status); and patient outcome.

OUTLINE:

Tumor DNA samples are examined by mutation analysis for germline and somatic mutations in the ALK tyrosine kinase domain. Samples are analyzed by whole genome amplification using polymerase chain reaction and then sequenced for DNA alterations in the entire ALK coding sequence. Samples are also examined for single nucleotide polymorphisms (SNPs) by polymorphism analysis. Exploratory multivariable analysis is performed to test for the prognostic ability of ALK mutations in the presence of other known prognostic variables (i.e., age, International Neuroblastoma Staging System stage, MYCN status, International Neuroblastoma Pathology Classification, and diploidy).

A subset of tumor DNA samples from high-risk patients will be resequenced for DNA alterations to determine whether or not additional regions in ALK, outside of the tyrosine kinase domain, are prone to mutations and should be sequenced in a larger panel.

ELIGIBILITY:
Inclusion Criteria:

* Tumor DNA samples available from pediatric patients with newly diagnosed neuroblastoma previously enrolled on clinical trial COG-ANBL00B1

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with newly diagnosed neuroblastoma previously enrolled on clinical trial COG-ANBL00B1.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2008-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to 1 year
  Using the log rank test, univariate comparisons of EFS and overall survival (OS) will be made for patients with ALK mutations versus those without ALK mutations.

SECONDARY OUTCOMES:
Overall survival | Up to 1 year
  Using the log rank test, univariate comparisons of EFS and OS will be made for patients with ALK mutations versus those without ALK mutations.
Disease progression as assessed by International Neuroblastoma Response Criteria | From the time of diagnosis until the time of first occurrence of relapse, progression, secondary malignancy, or death, or until the time of last contact if no event occurred, assessed up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yael Mosse, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States